CLINICAL TRIAL: NCT07151664
Title: Quality of Life Change in Patients Undergoing Parathyroidectomy With Secondary Hyperparathyroidism Due toEnd-stage Renal Failure: a Retrospective Cohort Study
Brief Title: Retrospective Analysis of Quality of Life Changes in Patients Undergoing Parathyroidectomy for End-Stage Renal Disease
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: 2024804
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Secondary Hyperparathyroidism Due to Renal Causes; End Stage Renal Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of life change in patients Undergoing Parathyroidectomy with end-stage renal failure: Quality of Life Progression in PatientsUndergoing Parathyroidectomy WithSecondary Hyperparathyroidism Due to End-stage Renal Failure
  Interventions: Other: Quality of life progression after parathyroidectomy

INTERVENTIONS:
Other: Quality of life progression after parathyroidectomy — Study the progression of quality of life

SUMMARY:
The purpose of this study is to characterize changes in quality of life in patients who had undergone parathyroidectomy for secondary hyperparathyroidism due to end-stage renal disease, based on data extracted from an established database

DETAILED DESCRIPTION:
Data were retrospectively collected from an established database of patients who underwent surgery for renal secondary hyperparathyroidism (SHPT). Extracted information included demographic and clinical characteristics (age, gender, education level, clinical symptoms), baseline quality of life assessed by the 36-item Short-Form Health Survey (SF-36), and completed follow-up assessments of SF-36 scores, depression, and anxiety at one, three, six months, and one year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years； Patients who had undergone parathyroidectomy for secondary hyperparathyroidism due to end-stage renal disease.

Exclusion Criteria:

Patients who underwent kidney transplantation during the study period. Patients with postoperative whole blood parathyroid hormone levels >300 pg/mL within the first week after surgery.

Patients with missing postoperative quality of life assessment data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had undergone parathyroidectomy for secondary hyperparathyroidism due to end-stage renal disease were included in this study
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Quality of life scores change with respect to time | up to 1 year
  Quality of life was assessed using the 36-item Short Form Health Survey (SF-36) scale. Completed responses for each of the 36 items were extracted from the database. Item responses were aggregated to calculate scores for each of the eight dimensions. Scores for each dimension range from 0 to 100, with higher scores indicating better health status

SECONDARY OUTCOMES:
Anxiety and depression score change with respect to time | up to 1 year
  Anxiety and depression were evaluated using the Hospital Anxiety and Depression Scale (HADS). Completed responses for the 14-item HADS, comprising 7 items each for the anxiety (HADS-A) and depression (HADS-D) subscales, were extracted from the database. Item scores range from 0 to 3, and were summed to yield separate scores for anxiety and depression
Bone pain scores change with respect to time | up to 1 year
  Bone pain was evaluated using the Numerical Rating Scale (NRS). Completed NRS scores, ranging from 0 to 10, were extracted from the database. In this scale, 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, 7-9 represents severe pain, and 10 represents the worst pain
Length of hospital stay | an average of 1 week

IPD SHARING:
Plan to Share IPD: No